CLINICAL TRIAL: NCT03218891
Title: Cardiac Rehabilitation in Patients With Refractory Angina
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Israelita Albert Einstein (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government); Instituto do Coracao (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014/00345-0
Record Dates: First submitted 2017-06-05; First posted 2017-07-17 (Actual); Last update posted 2022-02-11 (Actual); Status verified 2020-03

CONDITIONS: Refractory Angina
Keywords: Refractory Angina; Rehabilitation
MeSH Terms: conditions — Angina Pectoris | interventions — Cardiac Rehabilitation

STUDY DESIGN:
Intervention Model Description: 1. Optimized clinical treatment group + physical training for 12 weeks (TF);
  2. optimized clinical treatment group (CT);
  3. Group with coronary insufficiency without angina (CD);
  4. Group normal healthy subjects
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Clinical treatment physical training (Experimental): Patients with optimized clinical treatment group that will do physical training for 12 weeks. They will do the tests in moment 1 and after 3 mounths.
  The intervention is the Cardiac Rehabilitation.
  Interventions: Behavioral: Cardiac Rehabilitation
- Optimized clinical treatment (No Intervention): Patients with optimized clinical treatment group that will not do physical training.They will do the tests in moment 1 and after 3 mounths.
- Coronary insufficiency without angina (No Intervention): Group with coronary insufficiency without angina and will not do physical training. They will do the tests only one moment.
- Normal healthy subjects (No Intervention): Group normal healthy subjects, without coronary injuries, diabetes, hypertension and another chronic disease. These group have be sedentary and will not do physical training. They will do the tests only one moment.

INTERVENTIONS:
Behavioral: Cardiac Rehabilitation — The physical training program will start shortly after the initial exams have been completed. The physical training protocol will consist of a 12-week duration, with a frequency of 3 weekly sessions of 60 minutes duration each. The intensity will be prescribed from the echocardiogram with effort and cardiopulmonary test. All sessions will be monitored by telemetry and will be distributed as follows:
  * 5 minutes warm up
  * 30 to 40 minutes of aerobic exercise (treadmill). The training intensity will be prescribed individually, based on the results of the test results;
  * 10 minutes of localized exercises;
  * 5 minutes of relaxation.
  Arms: Clinical treatment physical training

SUMMARY:
The purpose of this study is to evaluate the safety and feasibility of cardiovascular rehabilitation in Patients with refractory angina, evaluate the effect of cardiovascular rehabilitation in patients with angina Refractory, by maximal oxygen consumption (VO2max) and global myocardial ischemic load by Stress Echocardiography; To evaluate the presence of myocardial injury, caused by physical stress, through ultra-sensitive troponin after sessions of aerobic physical activity, evaluating the behavior during the training period; To evaluate the effect of rehabilitation on the modulation of sympathetic activity and inflammation, muscular blood flow and lipid metabolism; To evaluate of the effect of rehabilitation on ventricular function through Stress echocardiography; Detection of ischemic episodes and arrhythmias identified during the Rehabilitation sessions through external cardiac monitoring (telemetry); Evaluate the quality of life assessment through the SF-36 questionnaire, Canadian Cardiovascular Society, the number of symptomatic episodes of ischemia, daily sublingual nitrate intake.

DETAILED DESCRIPTION:
After signing the informed consent form, patients will be randomized into 4 groups: 1. Optimized clinical treatment group + physical training for 12 weeks (TF); 2. optimized clinical treatment group (CT); 3. Group with coronary insufficiency without angina (CD); Group 4: normal healthy subjects All patients will be submitted to the following procedures in 2 moments * (times 0 and 3): -Routine laboratory tests including study of total cholesterol, LDL-cholesterol, -HDL-cholesterol, including study of the functionality of HDL-c, triglycerides, complete blood count, renal function, fasting glycemia, glycosylated hemoglobin (HbA1C); - Dosage of biomarkers of myocardial ischemia (ultra-sensitive troponin); - Dosage of inflammatory markers: Tumor necrosis factor (TNFn), interleukins 1 and 6 (IL-1 and IL-6), ultra-sensitive C-reactive protein (CRP); - Vascular endothelial growth factor (VEGF) dosage; - ergospirometric test in cycloergometer; - Echocardiogram with physical stress with evaluation of myocardial perfusion and function; - Evaluation of sympathetic activity through microneurography; - Evaluation of vascular reactivity through ultrasound of the brachial artery. - Evaluation of muscular blood flow through plethysmography; - Isometric exercise protocols; - Mental stress protocol - Quality of Life Questionnaire; - Diary of angina. After the initial examinations, the candidates of the TF group will be evaluated by cardiovascular rehabilitation team, for training prescription, which will be performed in a hospital environment, supervised by a qualified doctor. The rehabilitation may be interrupted in any patient, for safety measure, if the investigator deems it appropriate. All patients in both groups will receive clinical follow-up during the protocol, with monthly consultations during the 12-week protocol period (time 0 to 3), in which clinical evaluations of symptoms and quality of life of the patients will be performed . Any clinical intercurrence will be promptly annotated and evaluated according to the need of the moment. After this period, routine outpatient follow-up is scheduled at the outpatient clinic, and counseling for unsupervised physical training, according to the results of the study. All laboratory, clinical, imaging, and functional parameters will be evaluated before and at the end of the protocol.

ELIGIBILITY:
Group 1 and 2

Inclusion Criteria:

* Stable angina functional class II to IV according to the classification of Canadian Cardiovascular Society (CCS) 39, or limiting angina in Perception of the patient;
* Documented myocardial ischemia by imaging method;
* Patients not eligible for myocardial revascularization procedures surgical conventional, due to the unfavorable anatomy;
* Signature of the Free and Informed Consent Form.

Exclusion Criteria:

* Patients with definitive pacemaker or implantable cardioverter defibrillator (ICD);
* Patients with non-sinus heart rhythm;
* Patients with complete intraventricular block;
* Acute coronary syndrome (myocardial infarction or unstable angina) or previous procedures for myocardial revascularization (angioplasty / surgery) less than 3 months;
* Functional impossibility (orthopedic, rheumatic, neurological, or otherwise) or social for participation in the Rehabilitation Program;
* Classification of risk for American Heart Association class D physical training (unstable ischemia, stenosis or severe or symptomatic valve insufficiency, congenital heart disease, decompensated heart failure, uncontrolled arrhythmias and other conditions that may be aggravated by exercise).

Group 3

Inclusion Criteria:

* Patients with coronary insufficiency without angina;
* Signature of the Free and Informed Consent Form.

Group 4

Inclusion Criteria:

* Signature of the Free and Informed Consent Form;
* Healthy;
* Non-smokers;
* Sedentary

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2020-07-28 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Cardiovascular rehabilitation in patients with refractory angina is safe; | 3 months of rehabilitation
  Evaluated number of patients who have any kind of cardiovascular event during rehabilitation, as well as number of sore throat during the sessions.
Cardiovascular rehabilitation in patients with refractory angina is efficient; | 3 months of rehabilitation
  Evaluated number of sore throat during the sessions.
Improve the maximal oxygen consumption | 3 months of rehabilitation
  Improvement of Maximal oxygen uptake (VO2max)
Improve the global myocardial ischemic load | 3 months of rehabilitation
  Reduction of myocardial ischemia, evidenced by improvement of the standard by effort echocardiography

SECONDARY OUTCOMES:
Reduction of myocardial injury caused by physical stress | 3 months of rehabilitation
  Improves levels of Troponin-T after 1 exercise session at the initial moment of the Protocol and after 3 months.
Rehabilitation will modulate sympathetic activity | 3 months of rehabilitation
  Decreased sympathetic nerve activity measured by the amount of shots in his microneurography
Improvement of ventricular function | 3 months of rehabilitation
  Improvement of ventricular function through stress echocardiography in patients undergoing rehabilitation
Improvement of the quality of life | 3 months of rehabilitation
  Improvement of the quality of life measured through the SF-36 questionnaire.
Rehabilitation will increase muscle blood flow | 3 months of rehabilitation
  Increase peripheral muscle blood flow measured by plethysmography.
Reduction in the number of symptomatic episodes of ischemia | 3 months of rehabilitation
  Reduction in the number of episodes of ischemia, reduction of daily sublingual nitrate intake.
Reduction of the daily consumption of sublingual nitrate | 3 months of rehabilitation
  Reduction of daily sublingual nitrate intake.
Improve the functional class of Refractory Angina | 3 months of rehabilitation
  Improve the functional class decrease of angina (according to Canadian Cardiovascular Society classification)

CONTACTS AND LOCATIONS:
Overall Officials: Luciana Janot de Matos, Dra, Principal Investigator — Hospital Israelita Albert Einstein; Luciana Janot de Matos, Dra, Principal Investigator — InCor Heart Institute
Locations (1):
- Instituto Israelita de Ensino e Pesquisa Albert Einstein 's (IIEP), São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] de Assumpcao CRA, do Prado DML, Jordao CP, Dourado LOC, Vieira MLC, Montenegro CGSP, Negrao CE, Gowdak LHW, De Matos LDNJ. Cardiopulmonary exercise test in patients with refractory angina: functional and ischemic evaluation. Clinics (Sao Paulo). 2022 Feb 5;77:100003. doi: 10.1016/j.clinsp.2021.100003. eCollection 2022. PMID 35134662